CLINICAL TRIAL: NCT01220583
Title: A Randomized Phase II/Phase III Study of Adjuvant Concurrent Radiation and Chemotherapy Versus Radiation Alone in Resected High-Risk Malignant Salivary Gland Tumors
Brief Title: Radiation Therapy With or Without Chemotherapy in Treating Patients With High-Risk Malignant Salivary Gland Tumors That Have Been Removed By Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-1008; CDR0000686072; NCI-2013-00370
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer
Keywords: stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; high-grade salivary gland mucoepidermoid carcinoma; salivary gland adenocarcinoma; stage IVA salivary gland cancer; stage IVB salivary gland cancer; stage IVC salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms | interventions — Cisplatin; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients undergo 3-dimensional conformal radiotherapy (3D-CRT) or intensity-modulated radiotherapy (IMRT) 5 days a week for 6-6.5 weeks. Patients also receive cisplatin IV over 60 minutes on days 1, 8, 15, 22, 29, 36, and 43 during radiotherapy.
  Interventions: Drug: cisplatin; Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy
- Arm II (Experimental): Patients undergo 3D-CRT or IMRT as in arm I.
  Interventions: Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Drug: cisplatin — Given IV
  Arms: Arm I
Radiation: 3-dimensional conformal radiation therapy — Undergo radiotherapy
Radiation: intensity-modulated radiation therapy — Undergo radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether radiation therapy is more effective when given together with chemotherapy or alone after surgery in treating salivary gland tumors.

PURPOSE: This randomized phase II/III trial is studying radiation therapy with or without chemotherapy to see how well it works in treating patients with high-risk malignant salivary gland tumors that have been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

Phase II

* Determine the feasibility of conducting a cooperative group prospective clinical trial in patients with resected malignant salivary gland tumors.
* Acquire preliminary efficacy data comparing postoperative radiotherapy alone to concurrent chemotherapy and radiation using weekly cisplatin.

Phase III

* Compare overall survival rates among patients receiving cisplatin and radiation to those receiving radiation alone.

Secondary

Phase II/III

* Compare the acute toxicities of these 2 adjuvant treatments.
* Compare late treatment-related adverse events in patients receiving postoperative radiation to those receiving concurrent chemoradiation.
* Compare progression-free survival rates among patients receiving cisplatin and radiation to those receiving radiation alone in both the cohort of patients with pathologically high-risk disease (high-grade adenocarcinoma, high-grade mucoepidermoid carcinoma, salivary duct carcinoma), and the patient cohort with pathologically intermediate-risk disease (all other eligible diagnoses).
* Investigate quality of life and patient-reported outcomes in patients enrolled in the study.
* Identify the histopathology and tumor marker expression from patients enrolled on this trial and assemble a tissue bank for future correlative studies.
* Establish a NRG Oncology baseline database for salivary gland malignancies to serve as a resource for future exploration of innovative and/or targeted approaches for this disease.

OUTLINE: This is a multicenter study. Patients are stratified according to histology (high-grade mucoepidermoid carcinoma vs salivary duct carcinoma vs high-grade adenocarcinoma) and nodal status (N0 vs N1-3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo 3-dimensional conformal radiotherapy (3D-CRT) or intensity-modulated radiotherapy (IMRT) 5 days a week for 6-6.5 weeks. Patients also receive cisplatin IV over 60 minutes on days 1, 8, 15, 22, 29, 36, and 43 during radiotherapy.
* Arm II: Patients undergo 3D-CRT or IMRT as in Arm I. Tissue and blood samples may be collected for translational research studies. Patients may complete quality-of-life assessments periodically.

After completion of study treatment, patients are followed up at 3, 6, 9, 12, and 24 months, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically proven diagnosis of a malignant major salivary gland tumor or malignant minor salivary gland tumor of the head and neck of the following histologic subtypes:

  * Intermediate-grade adenocarcinoma or intermediate-grade mucoepidermoid carcinoma
  * High-grade acinic cell carcinoma or high-grade (>30% solid component) adenoid cystic carcinoma
* Surgical resection with curative intent within 8 weeks prior to registration
* All patients must have a Medical Oncology evaluation within 4 weeks prior to registration
* Pathologic stage T3-4 or N1-3 or T1-2, N0 with a close (≤ 1mm) or microscopically positive surgical margin; patients must be free of distant metastases based upon the following minimum diagnostic workup:

  * History/physical examination within 8 weeks prior to registration
  * Radiologic confirmation of the absence of hematogenous metastasis within 12 weeks prior to registration; at a minimum, contrast CT imaging of the chest is required (PET/CT is acceptable)
* No patients with residual macroscopic disease after surgery
* No prior systemic chemotherapy or radiation therapy for salivary gland malignancy

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute neutrophil count (ANC) ≥ 1,800 cells/mm^3
* Platelets ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 8.0 g/dL (the use of transfusion or other intervention to achieve hemoglobin ≥ 8.0 g/dL is acceptable)
* Serum creatinine < 2.0 mg/dL
* Total bilirubin < 2 x the institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x the institutional ULN
* Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential
* Women of childbearing potential and male participants who are sexually active must practice adequate contraception during treatment and for 6 weeks following treatment
* Not pregnant or nursing
* Patients must be deemed able to comply with the treatment plan and follow-up schedule
* Patients must provide study specific informed consent prior to study entry, including consent for mandatory tissue submission for central review
* No prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* No severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects (coagulation parameters are not required for entry into this protocol)
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition (HIV testing is not required for entry into this protocol)

    * Protocol-specific requirements may also exclude immunocompromised patients
  * Pre-existing ≥ grade 2 neuropathy
* No significant pre-existing hearing loss, as defined by the patient or treating physician

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy or radiation therapy for salivary gland malignancy (prior chemotherapy for a different cancer is allowable)
* No prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* No prior organ transplant
* No concurrent hematopoietic growth factors (e.g., G-CSF or pegfilgrastim) during radiotherapy
* No concurrent erythropoiesis-stimulating agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2011-01; Primary Completion 2026-10-31 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS), defined by the events of local-regional progression or recurrence, distant metastasis, or death from any cause, primarily at 2 years | From randomization to 2 years.

SECONDARY OUTCOMES:
Overall survival (OS) rate at 2 years | From randomization to 2 years.
PFS rate at 5 years | From randomization to 5 years.
OS rate at 5 years | From randomization to 5 years.
Treatment-related toxicity, defined as any grade 3-4 adverse events (CTCAE v. 4) deemed to be definitely, probably, or possibly related to protocol treatment | From start of treatment to last follow-up.
Treatment-related mortality, defined as any death during or within 30 days of discontinuation of protocol treatment | From start of treatment to 30 days after the end of treatment.
Chemotherapy delivery as measured by percentage of protocol prescription given | From start of treatment to end of treatment.
Radiation delivery as measured by elapsed treatment days | From start of treatment to end of treatment.
Determine whether quality of life, fatigue and xerostomia differ as a function of treatment assignment at 3, 12, and 24 months after completing radiotherapy. | From randomization to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina P. Rodriguez, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (268):
- United States (259):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - Arizona Breast Cancer Specialists-Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Arizona Breast Cancer Specialists-Phoenix, Phoenix, Arizona
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - Arizona Breast Cancer Specialists, Scottsdale, Arizona
  - Arizona Breast Cancer Specialists-Scottsdale, Scottsdale, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - William Backus Hospital, Norwich, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Saint Francis Hospital, Federal Way, Washington
  - Seattle Cancer Care Alliance at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (8):
  - Cross Cancer Institute, Edmonton, Alberta
  - Health Sciences North, Greater Sudbury, Ontario
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Joshi NP, Broughman JR. Postoperative Management of Salivary Gland Tumors. Curr Treat Options Oncol. 2021 Feb 9;22(3):23. doi: 10.1007/s11864-021-00820-9. PMID 33560478